CLINICAL TRIAL: NCT01204567
Title: The Aim of the Study is to Evaluate the Effect of Aerobic Fitness Training on Mental Health (Health-related Quality of Life), Cognitive and Physical Capacity in Older People Discharged From Hospital.
Brief Title: The Influence of Exercise on Mental Health After Discharge From Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/184a
Record Dates: First submitted 2010-09-10; First posted 2010-09-17 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Quality of Life
Keywords: HLRQ; elderly; aerobic fitness; cognitive capacity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training follow-up after discharge (Active Comparator): Aerobic training Home-program
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Aerobic training — Group-based Aerobic Interval Training twice a week in 12 weeks, based on the Ulleval model. The Norwegian Ulleval Model is a group-based aerobic interval training program which is widely used in Scandinavian hospitals for patients with coronary disease. It is designed to improve physical capacity, body awareness and emotional well-being.
  Other Names: 1 intervention group; 1 control group no follow-up

SUMMARY:
The aim of this study is to evaluate the effect of aerobic fitness training on mental health (health-related quality of life),cognitive and physical capacity in older people discharge from hospital and to assess if further aerobic training at home enhances the effect.

Design: Randomized controlled trial conducted at Oslo University Hospital, department of Medicine in conjunction with Oslo University College. The subjects will be randomized into one intervention group (training group) or one control group.

Outcome measure:

Health-related quality of life Physical function Cognitive capacity Physical activity Body composition Physical activity level

DETAILED DESCRIPTION:
Research has indicated that participation in a regular exercise program is an effective intervention to maintain and enhance cognitive and physical function in older individuals.Despite good evidence regarding the positive effects of exercise, a sedentary or inactive lifestyle is common among people over 65 years of old, especially among persons with chronic diseases. Research shows that good mental health and physical capacity is of vital importance for living independently in the community and we know that participation in physical activity offers good opportunities to extend years of active independent life. Nevertheless our knowledge is sparse regarding the evidence of effective programs for health promotion in groups of elderly, especially after discharge from hospital. Our knowledge is also sparse as to which intervention program is the most effective, group-based training or home- based training.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Be able to perform the Timed Up and Go test without use of assistive device

Exclusion Criteria:

* Chronic disease with expected lifespan < 1 year
* Exercise regularly more than twice a week
* Cognitive impairment MMS < 24
* Assessed by a doctor not to tolerate aerobic exercises
* Exercise limiting cardiovascular or musculoskeletal disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life. Short form Health Survey (SF-36, version 2 | 3 and 12 months

SECONDARY OUTCOMES:
Senior fitness test, Cognitive capacity, PASE | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Therese Brovold, phd student, Principal Investigator — no afflication
Locations (1):
- Oslo University Hospital, Oslo, Norway